CLINICAL TRIAL: NCT04668339
Title: A Phase 2 Randomized, Observer-Blind, Placebo-Controlled Study to Assess the Safety, Reactogenicity, and Immunogenicity of the SARS CoV-2 Vaccine ARCT-021 in Healthy Adult Participants
Brief Title: A Trial Evaluating the Safety and Effects of an RNA Vaccine ARCT-021 in Healthy Adults
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A decision was made to terminate the study for operational/business reasons. The study was not terminated for reasons of safety or immunogenicity.
Sponsor: Arcturus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ARCT-021-04
Record Dates: First submitted 2020-11-25; First posted 2020-12-16 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Covid19; SARS-CoV Infection; Corona Virus Infection
Keywords: SARS-CoV-2 Vaccine; Coronavirus Virus Diseases; RNA COVID 19; COVID 19 Vaccine Arcturus; self amplifying RNA vaccine
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: sequential assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Study Group 1, Younger Adult Participants (Experimental): Participants will receive one dose of ARCT-021 on Day 0, one dose of Placebo (saline) on Day 28 and on Day 208 either one dose of ARCT-021 or one dose of placebo
  Interventions: Biological: ARCT-021 single dose priming; Biological: Randomized booster
- Study Group 2, Younger Adult Participants (Experimental): Participants will receive one dose of ARCT-021 on Day 0, a second dose of ARCT-021 on Day 28 and on Day 208 either one dose of ARCT-021 or one dose of placebo
  Interventions: Biological: ARCT-021 two lower dose priming; Biological: Randomized booster
- Study Group 3, Younger Adult Participants (Experimental): Participants will receive one dose of ARCT-021 on Day 0, a second dose of ARCT-021 on Day 28 and on Day 208 either one dose of ARCT-021 or one dose of placebo
  Interventions: Biological: ARCT-021 two higher dose priming; Biological: Randomized booster
- Study Group 4, Younger Adult Participants (Placebo Comparator): Participants will receive one of Placebo (Saline) on Day 0, one dose of Placebo on Day 28, and one dose of Placebo on Day 208
  Interventions: Biological: Placebo (two doses), priming; Biological: Placebo booster
- Study Group 1, Older Adult Participants (Experimental): Participants will receive one dose of ARCT-021 on Day 0, one dose of Placebo (saline) on Day 28 and on Day 208 either one dose of ARCT-021 or one dose of placebo
  Interventions: Biological: ARCT-021 single dose priming; Biological: Randomized booster
- Study Group 2, Older Adult Participants (Experimental): Participants will receive one dose of ARCT-021 on Day 0, a second dose of ARCT-021 on Day 28 and on Day 208 either one dose of ARCT-021 or one dose of placebo
  Interventions: Biological: ARCT-021 two lower dose priming; Biological: Randomized booster
- Study Group 3, Older Adult Participants (Experimental): Participants will receive one dose of ARCT-021 on Day 0, a second dose of ARCT-021 on Day 28 and on Day 208 either one dose of ARCT-021 or one dose of placebo
  Interventions: Biological: ARCT-021 two higher dose priming; Biological: Randomized booster
- Study Group 4, Older Adult Participants (Placebo Comparator): Participants will receive one dose of Placebo (saline) on Day 0, a second dose of Placebo on Day 28 and a third dose of Placebo on Day 208
  Interventions: Biological: Placebo (two doses), priming; Biological: Placebo booster

INTERVENTIONS:
Biological: ARCT-021 single dose priming — ARCT-021 higher dose (one dose) + placebo (one dose)
  Arms: Study Group 1, Older Adult Participants; Study Group 1, Younger Adult Participants
Biological: ARCT-021 two lower dose priming — ARCT-021 lower dose (two doses, Day 0 and Day 28)
  Arms: Study Group 2, Older Adult Participants; Study Group 2, Younger Adult Participants
Biological: ARCT-021 two higher dose priming — ARCT-021 higher dose (two doses, Day 0 and Day 28)
  Arms: Study Group 3, Older Adult Participants; Study Group 3, Younger Adult Participants
Biological: Placebo (two doses), priming — Placebo (two doses, Day 0 and Day 28)
  Arms: Study Group 4, Older Adult Participants; Study Group 4, Younger Adult Participants
Biological: Randomized booster — ARCT-021 (single dose) OR placebo, booster
  Arms: Study Group 1, Older Adult Participants; Study Group 1, Younger Adult Participants; Study Group 2, Older Adult Participants; Study Group 2, Younger Adult Participants; Study Group 3, Older Adult Participants; Study Group 3, Younger Adult Participants
Biological: Placebo booster — Placebo (single dose)
  Arms: Study Group 4, Older Adult Participants; Study Group 4, Younger Adult Participants

SUMMARY:
This is a Phase 2, randomized, placebo-controlled, and observer-blind study in healthy adults.

The study will evaluate the safety, tolerability, and immunogenicity of the SARS-CoV-2 RNA vaccine candidate against COVID-19:

As 2 doses (at two different dose levels), separated by 28 days or as 1 dose

In adults 18 years of age and older

DETAILED DESCRIPTION:
This is a multiregional, multicenter, Phase 2, randomized, observer-blind study designed to evaluate the safety, reactogenicity, and immunogenicity of the study vaccine in younger and older adult participants. Enrolled participants will be randomly assigned to receive either study vaccine ARCT-021 or placebo (sterile saline).

Approximately 600 participants (300 each in younger [18 to <56 years of age in United States or 21 to <56 years of age in Singapore] and older [≥56 years of age] participants) will be enrolled (including at least 50% of participants in the older cohort ≥65 years of age). Participants will be stratified by age and then randomly assigned (3 ARCT-021:1 placebo) to receive 2 doses of study vaccine separated by 28 days. At 180 days after second study vaccination (Day 208), participants in Study Groups 1, 2, and 3 will be randomly assigned again to receive a single booster dose of study vaccine (randomly assigned as 1 ARCT-021:1 placebo). Study Group 4 will not be randomized but will receive 1 dose of placebo at Day 208. Study Groups are summarized in Table 1. Study vaccine will be administered in an observer-blind fashion. Participants will be followed for safety and immunogenicity through 180 days after booster vaccination (Day 388). At a subset of clinical sites, all enrolled participants will also undergo blood sampling for evaluation of CMI responses.

Vaccine doses will be assigned as follows:

Younger Age Cohort:

Study Group 1: n= 75 participants, ARCT-021 7.5 µg (first dose), Placebo (second dose Study Group 2: n= 75 participants, ARCT-021 5.0 µg (first dose), 5.0 µg (second dose) Study Group 3: n= 75 participants, ARCT-021 7.5 µg (first dose), 7.5 µg (second dose) Study Group 4: n= 75 participants, Placebo (first dose), Placebo (second dose)

Booster Vaccine:

Study Groups 1, 2, 3: 113 participants, ARCT-021 5.0 µg or 7.5 µg, 112 participants, Placebo Study Group 4: n= 75 participants, Placebo

Older Age Cohort:

Study Group 1: n= 75 participants, ARCT-021 7.5 µg (first dose), Placebo (second dose Study Group 2: n= 75 participants, ARCT-021 5.0 µg (first dose), 5.0 µg (second dose) Study Group 3: n= 75 participants, ARCT-021 7.5 µg (first dose), 7.5 µg (second dose) Study Group 4: n= 75 participants, Placebo (first dose), Placebo (second dose)

Booster Vaccine:

Study Groups 1, 2, 3: 113 participants, ARCT-021 5.0 µg or 7.5 µg, 112 participants, Placebo Study Group 4: n= 75 participants, Placebo

A DSMB will be in place to independently review the safety data of participants. Pausing Rules are also utilized in this study to reduce risk to study participants.

The expected duration of participation for an individual participant is approximately 14 months, inclusive of the Screening period.

ELIGIBILITY:
Inclusion Criteria:

Individuals who:

1. are able to provide consent
2. agree to comply with all study visits and procedures
3. are willing and able to adhere to study restrictions
4. are sexually active and willing to adhere to contraceptive requirements
5. are male or female ≥18 or (in Singapore) ≥21 years of age
6. are medically stable

Exclusion Criteria:

Individuals who:

1. have had SARS-CoV-2 infection or COVID-19 disease.
2. have had cancer except for cancers that were treated and that have low risk of returning
3. have chronic kidney disease
4. have some chronic lung diseases
5. have some heart conditions
6. have compromised immune systems
7. are obese
8. have sickle cell disease or some other blood disorders
9. are current smokers and/or use illegal drugs
10. have Type 2 diabetics
11. are immunocompromised, immunodeficient or have had a transplant
12. have autoimmune disease
13. have other severe or uncontrolled diseases or disease that may interfere with the interpretation of the study
14. have a positive test for hepatitis B or C or human immunodeficiency virus
15. have had a severe reaction to previous investigational vaccines
16. have a fever or are feeling sick close to the time of the first vaccination of the study
17. have positive drug test at screening
18. are pregnant
19. are breastfeeding
20. have a bleeding disorder
21. have previously received an investigational coronavirus vaccine (SARS-CoV(1) or MERS) or who plan to be in other COVID-19 studies
22. have recently been vaccinated with other vaccines
23. have recently received blood products
24. who work at one of the clinic sites participating in this study, work at Arcturus, who work at other companies that monitor the study or close family members to the sites, Arcturus, or partners involved in study monitoring
25. other restrictions may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 581 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (12):
  - Arcturus Investigational Site 103, Chandler, Arizona
  - Arcturus Investigational Site 107, Tucson, Arizona
  - Arcturus Investigational Site 112, San Diego, California
  - Arcturus Investigational Site 104, Melbourne, Florida
  - Arcturus Investigational Site 105, Orlando, Florida
  - Arcturus Investigational Site 106, Pinellas Park, Florida
  - Arcturus Investigational Site 109, The Villages, Florida
  - Arcturus Investigational Site 101, Peoria, Illinois
  - Arcturus Investigational Site 110, Rockville, Maryland
  - Arcturus Investigational Site 102, Anderson, South Carolina
  - Arcturus Investigational Site 111, Austin, Texas
  - Arcturus Investigational Site 108, Dallas, Texas
- Singapore (3):
  - Arcturus Investigational Site 204, Singapore
  - Arcturus Investigational Site 201, Singapore
  - Arcturus Investigational Site 203, Singapore

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be made available to study investigators at this time.

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment A: Participants in this group received ARCT-021 7.5 micrograms (mcg) at Day 0 and placebo matched to ARCT-021 at Day 28. Participants who did not otherwise have any contraindications to additional study vaccinations were randomly assigned to ARCT-021, ARCT-154, ARCT-165, or placebo for a third (booster) dose of study vaccine given at Day 208.
- Treatment B: Participants in this group received ARCT-021 5 mcg at Day 0 and ARCT-021 5 mcg at Day 28. Participants who did not otherwise have any contraindications to additional study vaccinations were randomly assigned to ARCT-021, ARCT-154, ARCT-165, or placebo for a third (booster) dose of study vaccine given at Day 208.
- Treatment C: Participants in this group received ARCT-021 7.5 mcg at Day 0 and ARCT-021 7.5 mcg at Day 28. Participants who did not otherwise have any contraindications to additional study vaccinations were randomly assigned to ARCT-021, ARCT-154, ARCT-165, or placebo for a third (booster) dose of study vaccine given at Day 208.
- Treatment D: Participants in this group received placebo matched to ARCT-021 at Day 0 and placebo matched to ARCT-021 at Day 28. Participants who did not otherwise have any contraindications to additional study vaccinations were randomly assigned to ARCT-021, ARCT-154, ARCT-165, or placebo for a third (booster) dose of study vaccine given at Day 208.
Period: Overall Study
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Started | 146 | 145 | 145 | 145
Received Vaccination 1 | 146 | 145 | 144 | 145
Received Vaccination 2 | 132 | 135 | 139 | 139
Received Booster Vaccination | 51 | 60 | 58 | 1
Booster - ARCT-021 5 mcg | 13 | 16 | 15 | 0
Booster - ARCT-154 5 mcg | 12 | 15 | 14 | 0
Booster - ARCT-165 5 mcg | 14 | 14 | 14 | 0
Booster - Placebo | 12 | 14 | 15 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 146 | 145 | 145 | 145
Not completed — Physician Decision | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 14 | 12 | 8 | 5
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Other than specified | 3 | 0 | 1 | 0
Not completed — Participant unblinded between Day 98 and 198 | 6 | 5 | 4 | 91
Not completed — Vaccine not Administered | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 18 | 23 | 12 | 20
Not completed — Withdrawal by Subject | 45 | 46 | 46 | 27
Not completed — Study Terminated by Sponsor | 59 | 59 | 71 | 1

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who received at least 1 dose of priming study vaccine (ARCT-021 or placebo). Participants were analyzed according to the vaccine received at the time of priming or booster vaccination. One participant who was randomized to group A received treatment dosing and schedule for group D due to a dosing error. This participant is included in group D for the safety set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Total
Number analyzed (Participants) | 145 | 144 | 145 | 146 | 580
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (16.15) | 49.9 (15.16) | 48.2 (17.08) | 48.2 (15.59) | 48.8 (15.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 71 | 60 | 65 | 266
  Male | 75 | 73 | 85 | 81 | 314
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 22 | 22 | 12 | 70
  Not Hispanic or Latino | 131 | 121 | 123 | 134 | 509
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 1 | 3
  Asian | 28 | 23 | 19 | 23 | 93
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 7 | 8 | 15 | 34
  White | 108 | 107 | 109 | 105 | 429
  More than one race | 1 | 2 | 3 | 1 | 7
  Unknown or Not Reported | 4 | 3 | 6 | 1 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Solicited Local Adverse Events Within 7 Days Post Each Priming Vaccination
Description: Per prespecified analysis, solicited local adverse events were defined as pain, erythema, swelling, or injection site tenderness. Solicited adverse reactions were recorded by the participant in an eDiary. Per prespecified analysis, solicited adverse events were not evaluated for severity (such as, serious or non-serious). A summary of all unsolicited adverse events and solicited adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: For 7 days following each dose administration (Day 0 up to Day 7 for Vaccination 1 and Day 29 up to Day 35 for Vaccination 2)
Population: The Reactogenicity analysis set included all participants who received any dose of priming study vaccine (ARCT-021 or placebo) and provided at least 1 reactogenicity diary report for the time period evaluated. Here, number analyzed signifies those participants who were evaluable in specified categories only.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 142 | 142 | 144 | 146
percentage of participants
  Vaccination 1: Pain | 52.8 | 48.6 | 57.6 | 8.2
  Vaccination 1: Erythema (Redness) | 14.8 | 19.7 | 11.1 | 7.5
  Vaccination 1: Swelling (Hardness) | 11.3 | 15.5 | 9.0 | 5.5
  Vaccination 1: Injection Site Tenderness | 79.6 | 75.4 | 83.3 | 19.9
  Vaccination 2: Pain: number analyzed (Participants) | 127 | 130 | 137 | 134
  Vaccination 2: Pain | 7.9 | 33.1 | 44.5 | 5.9
  Vaccination 2: Erythema (Redness): number analyzed (Participants) | 127 | 130 | 137 | 134
  Vaccination 2: Erythema (Redness) | 7.1 | 14.6 | 8.0 | 8.9
  Vaccination 2: Swelling (Hardness): number analyzed (Participants) | 127 | 130 | 137 | 134
  Vaccination 2: Swelling (Hardness) | 4.7 | 11.5 | 4.4 | 3.0
  Vaccination 2: Injection Site Tenderness: number analyzed (Participants) | 127 | 130 | 137 | 134
  Vaccination 2: Injection Site Tenderness | 15.0 | 67.7 | 75.2 | 15.6

2. Primary Outcome: Percentage of Participants Reporting Solicited Local Adverse Events Within 7 Days Post Booster Vaccination
Description: as for outcome 1
Time Frame: For 7 days following each dose administration (Day 208 up to Day 215)
Population: The Booster Reactogenicity analysis set included all participants who received any dose of booster vaccination (ARCT-021, ARCT-145, ARCT-156 or placebo) and provided at least 1 diary entry for the time period evaluated. Participants were analyzed according to the vaccine actually received. Here, overall number of participants analyzed signifies those who were evaluable for this outcome measure and number analyzed signifies those participants who were evaluable in specified categories only.
Measure: Number; unit: percentage of participants
Groups:
- Treatment E1: Participants in this group received booster dose of ARCT-021 5 mcg at Day 208.
- Treatment F1: Participants in this group received booster dose of ARCT-154 5 mcg at Day 208.
- Treatment G1: Participants in this group received booster dose of ARCT-165 5 mcg at Day 208.
- Treatment H1: Participants in this group received placebo at Day 208.
Arm/Group | Treatment E1 | Treatment F1 | Treatment G1 | Treatment H1
Number analyzed (Participants) | 41 | 36 | 38 | 39
percentage of participants
  Pain | 51.2 | 36.8 | 39.5 | 5.1
  Erythema (Redness) | 9.3 | 7.9 | 7.9 | 2.6
  Swelling (Hardness) | 11.6 | 5.3 | 7.9 | 0
  Injection Site Tenderness | 81.4 | 65.8 | 73.7 | 12.8

3. Primary Outcome: Percentage of Participants Reporting Solicited Systemic Adverse Events Within 7 Days Post Each Priming Vaccination
Description: Per prespecified analysis, solicited systemic adverse events were defined as fever, headache, fatigue, myalgia, arthralgia, nausea, chills, diarrhea, dizziness, and vomiting. Per prespecified analysis, solicited adverse events were not evaluated for severity (such as, serious or non-serious). A summary of all unsolicited adverse events and solicited adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 142 | 142 | 144 | 146
percentage of participants
  Vaccination 1: Fever: number analyzed (Participants) | 142 | 142 | 143 | 146
  Vaccination 1: Fever | 4.2 | 2.1 | 2.8 | 0
  Vaccination 1: Headache | 43.0 | 34.5 | 39.6 | 19.2
  Vaccination 1: Fatigue: number analyzed (Participants) | 142 | 142 | 144 | 145
  Vaccination 1: Fatigue | 47.2 | 36.6 | 40.3 | 20.5
  Vaccination 1: Myalgia: number analyzed (Participants) | 142 | 142 | 144 | 145
  Vaccination 1: Myalgia | 44.4 | 28.9 | 39.6 | 8.2
  Vaccination 1: Arthralgia: number analyzed (Participants) | 142 | 142 | 144 | 145
  Vaccination 1: Arthralgia | 21.1 | 15.5 | 17.4 | 8.2
  Vaccination 1: Nausea: number analyzed (Participants) | 142 | 142 | 144 | 145
  Vaccination 1: Nausea | 10.6 | 8.5 | 6.3 | 7.5
  Vaccination 1: Chills: number analyzed (Participants) | 142 | 142 | 144 | 145
  Vaccination 1: Chills | 28.9 | 16.9 | 22.9 | 2.1
  Vaccination 1: Diarrhea: number analyzed (Participants) | 142 | 142 | 144 | 145
  Vaccination 1: Diarrhea | 12.0 | 12.7 | 16.0 | 9.6
  Vaccination 1: Dizziness: number analyzed (Participants) | 142 | 142 | 144 | 145
  Vaccination 1: Dizziness | 7.7 | 9.9 | 9.0 | 8.9
  Vaccination 1: Vomiting: number analyzed (Participants) | 142 | 142 | 144 | 145
  Vaccination 1: Vomiting | 1.4 | 0 | 0 | 0
  Vaccination 2: Fever: number analyzed (Participants) | 123 | 129 | 131 | 134
  Vaccination 2: Fever | 0.8 | 3.1 | 6.6 | 0
  Vaccination 2: Headache: number analyzed (Participants) | 127 | 130 | 136 | 135
  Vaccination 2: Headache | 12.6 | 30.0 | 40.9 | 16.3
  Vaccination 2: Fatigue: number analyzed (Participants) | 127 | 130 | 136 | 135
  Vaccination 2: Fatigue | 14.2 | 33.1 | 44.5 | 21.5
  Vaccination 2: Myalgia: number analyzed (Participants) | 127 | 130 | 136 | 135
  Vaccination 2: Myalgia | 6.3 | 34.6 | 32.8 | 14.1
  Vaccination 2: Arthralgia: number analyzed (Participants) | 127 | 130 | 136 | 135
  Vaccination 2: Arthralgia | 3.1 | 16.9 | 24.1 | 9.6
  Vaccination 2: Nausea: number analyzed (Participants) | 127 | 130 | 136 | 135
  Vaccination 2: Nausea | 5.5 | 6.9 | 8.8 | 5.2
  Vaccination 2: Chills: number analyzed (Participants) | 127 | 130 | 136 | 135
  Vaccination 2: Chills | 2.4 | 13.1 | 22.6 | 5.2
  Vaccination 2: Diarrhea: number analyzed (Participants) | 127 | 130 | 136 | 135
  Vaccination 2: Diarrhea | 7.1 | 10.0 | 10.9 | 12.6
  Vaccination 2: Dizziness: number analyzed (Participants) | 127 | 130 | 136 | 135
  Vaccination 2: Dizziness | 7.1 | 4.6 | 17.5 | 6.7
  Vaccination 2: Vomiting: number analyzed (Participants) | 127 | 130 | 136 | 135
  Vaccination 2: Vomiting | 0 | 0 | 0 | 0.7

4. Primary Outcome: Percentage of Participants Reporting Solicited Systemic Adverse Events Within 7 Days Post Booster Vaccination
Description: as for outcome 3
Time Frame: For 7 days post booster dose administration (Day 208 up to Day 215)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Treatment E1 | Treatment F1 | Treatment G1 | Treatment H1
Number analyzed (Participants) | 41 | 35 | 38 | 38
percentage of participants
  Fever: number analyzed (Participants) | 40 | 34 | 37 | 37
  Fever | 11.6 | 0 | 5.3 | 2.6
  Headache | 60.5 | 34.2 | 31.6 | 25.6
  Fatigue | 69.8 | 34.2 | 50.0 | 25.6
  Myalgia | 62.8 | 31.6 | 42.1 | 12.8
  Arthralgia | 48.8 | 21.1 | 31.6 | 12.8
  Nausea | 27.9 | 7.9 | 10.5 | 2.6
  Chills | 44.2 | 18.4 | 21.1 | 7.7
  Diarrhea | 25.6 | 18.4 | 10.5 | 10.3
  Dizziness | 32.6 | 10.5 | 10.5 | 2.6
  Vomiting | 7.0 | 2.6 | 0 | 0

5. Primary Outcome: Percentage of Participants Reporting Unsolicited Adverse Events Up to 28 Days Post Each Priming Vaccination
Description: An unsolicited AE was defined as any AE (serious and nonserious) occurring after administration of first dose of study vaccine and before the end of study. A summary of all unsolicited adverse events and solicited adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: 28 days following each dose administration (Day 0 up to Day 28 for Vaccination 1 and Day 29 up to Day 56 for Vaccination 2)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 145 | 144 | 145 | 146
percentage of participants
  Vaccination 1 | 20.7 | 22.2 | 17.9 | 19.2
  Vaccination 2: number analyzed (Participants) | 131 | 134 | 140 | 140
  Vaccination 2 | 19.1 | 19.4 | 8.6 | 20.7

6. Primary Outcome: Percentage of Participants Reporting Unsolicited Adverse Events Up to 28 Days Post Booster Vaccination
Description: as for outcome 5
Time Frame: 28 days following each dose administration (Day 208 up to 236 days)
Population: Booster Safety Set included all participants who received at least 1 dose of booster study vaccine (ARCT-021, ARCT-154, ARCT-165, or placebo) or had safety data collected in the period following booster administration.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment E1 | Treatment F1 | Treatment G1 | Treatment H1
Number analyzed (Participants) | 44 | 41 | 42 | 99
percentage of participants | 15.9 | 14.6 | 11.9 | 9.1

7. Primary Outcome: Percentage of Participants Reporting Treatment-Emergent Serious Adverse Events (SAE), Medically Attended Adverse Events (MAAE) and New Onset of Chronic Disease (NOCD) Post Each Priming Vaccination
Description: SAEs were defined as any event that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, resulted in a congenital anomaly or birth defect, or was an important medical event. An NOCD was defined as any AE that led to the new diagnosis of a chronic medical condition that was not present or suspected prior to enrollment. An MAAE was an AE that led to an unscheduled visit (including a telemedicine visit) to a healthcare practitioner. A summary of all unsolicited adverse events and solicited adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Up to Day 207
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 145 | 144 | 145 | 146
percentage of participants
  Any SAEs | 0 | 2.1 | 0.7 | 2.1
  Any MAAEs | 16.6 | 20.8 | 18.6 | 17.1
  Any NOCDs | 4.1 | 7.6 | 2.8 | 2.7

8. Primary Outcome: Percentage of Participants Reporting Treatment-emergent Serious Adverse Events, Medically Attended Adverse Events and New Onset of Chronic Disease Post Booster Vaccination
Description: SAEs were defined as any event that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, resulted in a congenital anomaly or birth defect, or was an important medical event. An NOCD was defined as an AE that led to the new diagnosis of a chronic medical condition that was not present or suspected prior to enrollment. An MAAE was an AE that led to an unscheduled visit (including a telemedicine visit) to a healthcare practitioner. A summary of all unsolicited adverse events and solicited adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Day 208 to early termination (up to 396 days)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Treatment E1 | Treatment F1 | Treatment G1 | Treatment H1
Number analyzed (Participants) | 44 | 41 | 42 | 99
percentage of participants
  Any SAEs | 0 | 0 | 2.4 | 0
  Any MAAEs | 11.4 | 19.5 | 11.9 | 12.1
  Any NOCDs | 2.3 | 4.9 | 0 | 0

9. Primary Outcome: Geometric Mean Titer (GMT) of Serum Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Neutralizing Antibodies Post Priming Vaccination
Time Frame: Day 1
Population: Modified intent to treat (mITT) analysis set included all participants who received at least 1 dose of study vaccine and who had pre- and post-vaccination immunogenicity data evaluable by the assay in use with valid results for the relevant time point. The mITT analysis set was analyzed according to vaccine received. Here, overall number of participants analyzed signifies those who were evaluable for this outcome measure only.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 131 | 140 | 134 | 141
IU/mL | 4.40 [4.03 to 4.80] | 5.14 [4.47 to 5.90] | 5.31 [4.57 to 6.18] | 4.75 [4.30 to 5.25]

10. Primary Outcome: GMT of SARS-CoV-2 Neutralizing Antibodies Post Priming Vaccination
Time Frame: Day 56
Population: mITT Analysis Set included all participants who received at least 1 dose of study vaccine and who had pre- and post-vaccination immunogenicity data evaluable by the assay in use with valid results for the relevant time point. The mITT analysis set was analyzed according to vaccine received. Here, overall number of participants analyzed signifies those who were evaluable for this outcome measure only.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 114 | 116 | 117 | 116
Titer | 5.47 [4.61 to 6.48] | 13.37 [10.65 to 16.79] | 15.31 [11.89 to 19.72] | 4.21 [3.89 to 4.57]

11. Primary Outcome: GMT of SARS-CoV-2 Neutralizing Antibodies Post Booster Vaccination
Time Frame: Day 208
Population: Booster mITT Analysis Set included all mITT participants who had at least 1 immunogenicity data evaluable by the assay in use with valid results during the booster vaccination period. Here, overall number of participants analyzed signifies those who were evaluable for this outcome measure only.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Treatment E1 | Treatment F1 | Treatment G1 | Treatment H1
Number analyzed (Participants) | 41 | 35 | 37 | 49
Titer | 13.37 [7.84 to 22.80] | 20.71 [10.47 to 40.97] | 14.04 [7.14 to 27.62] | 11.84 [7.57 to 18.51]

12. Primary Outcome: GMT of SARS-CoV-2 Neutralizing Antibodies Post Booster Vaccination
Time Frame: Day 236
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Treatment E1 | Treatment F1 | Treatment G1 | Treatment H1
Number analyzed (Participants) | 40 | 35 | 35 | 34
Titer | 229.70 [135.70 to 388.80] | 503.18 [296.57 to 853.72] | 380.77 [249.24 to 581.71] | 10.73 [6.56 to 17.56]

13. Primary Outcome: Geometric Mean Fold Rise (GMFR) in SARS-CoV-2 Neutralizing Antibody Titers Post Priming Vaccination
Description: GMFR is reported as a ratio to baseline (Day 0).
Time Frame: Day 56
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 114 | 116 | 117 | 116
Ratio | 1.3 [1.1 to 1.6] | 2.7 [2.2 to 3.5] | 2.9 [2.2 to 3.7] | 0.9 [0.8 to 1.0]

14. Primary Outcome: Geometric Mean Fold Rise (GMFR) in SARS-CoV-2 Neutralizing Antibody Titers Post Booster Vaccination
Description: GMFR is reported as a ratio to baseline (Day 0).
Time Frame: Day 208
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Treatment E1 | Treatment F1 | Treatment G1 | Treatment H1
Number analyzed (Participants) | 41 | 35 | 37 | 49
Ratio | 2.4 [1.3 to 4.6] | 4.2 [2.1 to 8.3] | 3.0 [1.6 to 5.7] | 2.0 [1.5 to 2.8]

15. Primary Outcome: GMFR in SARS-CoV-2 Neutralizing Antibody Titers Post Booster Vaccination
Description: GMFR is reported as a ratio to baseline (Day 0).
Time Frame: Day 236
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Treatment E1 | Treatment F1 | Treatment G1 | Treatment H1
Number analyzed (Participants) | 40 | 35 | 35 | 34
Ratio | 41.3 [22.0 to 77.7] | 100.8 [59.6 to 170.5] | 86.1 [58.8 to 126.1] | 1.7 [1.3 to 2.1]

16. Primary Outcome: Percentages of Participants Achieving Greater Than or Equal to 2-fold and 4-fold Increase From Before Vaccination (Baseline) in SARS-CoV-2 Serum Neutralizing Antibody Levels at Day 56
Time Frame: Baseline up to Day 56
Population: mITT analysis set included all participants who received at least 1 dose of study vaccine and who had pre- and post-vaccination immunogenicity data evaluable by the assay in use with valid results for the relevant time point. Here, overall number of participants analyzed signifies those who were evaluable for this outcome measure only.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 114 | 116 | 117 | 116
percentage of participants
  >=2-fold Increase from Baseline | 15.8 | 59.5 | 62.4 | 2.6
  >=4-fold Increase from Baseline | 8.8 | 43.1 | 42.7 | 0.9

17. Primary Outcome: Percentages of Participants Achieving Greater Than or Equal to 2-fold and 4-fold Increase From Before Vaccination (Baseline) in SARS-CoV-2 Serum Neutralizing Antibody Levels at Day 208
Time Frame: Baseline up to Day 208
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Treatment E1 | Treatment F1 | Treatment G1 | Treatment H1
Number analyzed (Participants) | 41 | 35 | 37 | 49
percentage of participants
  >=2-fold Increase from Baseline | 53.7 | 74.3 | 48.6 | 53.1
  >=4-fold Increase from Baseline | 26.8 | 25.7 | 21.6 | 14.3

18. Primary Outcome: Percentages of Participants Achieving Greater Than or Equal to 2-fold and 4-fold Increase From Before Vaccination (Baseline) in SARS-CoV-2 Serum Neutralizing Antibody Levels at Day 236
Time Frame: Baseline up to Day 236
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Treatment E1 | Treatment F1 | Treatment G1 | Treatment H1
Number analyzed (Participants) | 40 | 35 | 35 | 34
percentage of participants
  >=2-fold Increase from Baseline | 90.0 | 97.1 | 100 | 50.0
  >=4-fold Increase from Baseline | 85.0 | 94.3 | 100 | 8.8

19. Secondary Outcome: Geometric Mean Concentration of SARS-CoV-2 Anti-S1, Anti-RBD, and Anti-N Binding Antibody Levels Post Priming Vaccination
Time Frame: Days 0 and 56
Population: mITT analysis set included all participants who received at least 1 dose of study vaccine and who had pre- and post-vaccination immunogenicity data evaluable by the assay in use with valid results for the relevant time point. Here, overall number of participants analyzed signifies those who were evaluable for this outcome measure only and number analyzed signifies those participants who were evaluable at specified time points only.
Measure: Geometric Mean (95% Confidence Interval); unit: Binding antibody units/milliliters
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 131 | 140 | 133 | 141
Binding antibody units/milliliters
  Anti-N: Day 0 | 0.27 [0.21 to 0.35] | 0.26 [0.20 to 0.33] | 0.29 [0.22 to 0.37] | 0.29 [0.22 to 0.38]
  Anti-N: Day 56: number analyzed (Participants) | 114 | 115 | 117 | 116
  Anti-N: Day 56 | 0.23 [0.17 to 0.30] | 0.22 [0.17 to 0.30] | 0.27 [0.20 to 0.36] | 0.23 [0.17 to 0.31]
  Anti-RBD: Day 0 | 0.63 [0.50 to 0.80] | 0.58 [0.46 to 0.72] | 0.70 [0.53 to 0.93] | 0.56 [0.46 to 0.67]
  Anti-RBD: Day 56: number analyzed (Participants) | 114 | 115 | 117 | 116
  Anti-RBD: Day 56 | 5.19 [3.85 to 7.01] | 22.94 [17.25 to 30.51] | 35.71 [26.33 to 48.42] | 0.55 [0.43 to 0.71]
  Anti-S1: Day 0 | 0.40 [0.32 to 0.50] | 0.41 [0.33 to 0.51] | 0.53 [0.40 to 0.71] | 0.35 [0.28 to 0.42]
  Anti-S1: Day 56: number analyzed (Participants) | 114 | 115 | 117 | 116
  Anti-S1: Day 56 | 7.61 [5.93 to 9.78] | 25.91 [20.02 to 33.54] | 41.36 [32.59 to 52.49] | 0.34 [0.26 to 0.44]

20. Secondary Outcome: Geometric Mean Concentration of SARS-CoV-2 Anti-S1, Anti-RBD, and Anti-N Binding Antibody Levels Post Booster Vaccination
Time Frame: Day 208 and 236
Population: Booster mITT Analysis Set included all mITT participants who had at least 1 immunogenicity data evaluable by the assay in use with valid results during the booster vaccination period. Here, overall number of participants analyzed signifies those who were evaluable for this outcome measure only and number analyzed signifies those participants who were evaluable at specified time points only.
Measure: Geometric Mean (95% Confidence Interval); unit: Binding antibody units/milliliters
Arm/Group | Treatment E1 | Treatment F1 | Treatment G1 | Treatment H1
Number analyzed (Participants) | 41 | 35 | 36 | 49
Binding antibody units/milliliters
  Anti- N: Day 208 | 0.39 [0.22 to 0.66] | 0.38 [0.22 to 0.66] | 0.43 [0.23 to 0.79] | 0.40 [0.24 to 0.67]
  Anti-N: Day 236: number analyzed (Participants) | 40 | 35 | 35 | 34
  Anti-N: Day 236 | 0.67 [0.41 to 1.10] | 0.54 [0.34 to 0.85] | 0.73 [0.45 to 1.21] | 0.32 [0.18 to 0.58]
  Anti- S1: Day 208 | 10.10 [5.42 to 18.82] | 17.22 [7.85 to 37.77] | 13.36 [6.44 to 27.72] | 9.13 [5.21 to 15.99]
  Anti- S1: Day 236: number analyzed (Participants) | 40 | 35 | 35 | 34
  Anti- S1: Day 236 | 236.46 [144.96 to 385.74] | 488.81 [284.81 to 838.92] | 441.16 [316.21 to 615.48] | 5.97 [3.11 to 11.46]
  Anti- RBD: Day 208 | 10.29 [5.33 to 19.84] | 17.31 [7.23 to 41.42] | 12.81 [5.66 to 29.02] | 8.81 [4.73 to 16.41]
  Anti- RBD: Day 236: number analyzed (Participants) | 40 | 35 | 35 | 34
  Anti- RBD: Day 236 | 258.97 [140.12 to 478.63] | 715.15 [394.23 to 1297.31] | 591.87 [397.34 to 881.64] | 5.38 [2.63 to 11.01]

21. Secondary Outcome: Geometric Mean Fold Rise (GMFR) in SARS-CoV-2 Anti-S1, Anti-RBD, and Anti-N Binding Antibody Levels Before Vaccination to Day 56
Time Frame: Day 56
Population: as for outcome 16
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 114 | 115 | 117 | 116
Ratio
  Anti-N | 0.9 [0.8 to 0.9] | 0.9 [0.8 to 1.0] | 0.9 [0.8 to 1.0] | 0.9 [0.9 to 1.0]
  Anti-RBD | 8.6 [6.3 to 11.8] | 42.7 [32.0 to 57.0] | 48.7 [34.3 to 69.3] | 1.0 [0.9 to 1.1]
  Anti-S1 | 19.8 [14.8 to 26.4] | 65.9 [50.3 to 86.5] | 77.7 [55.2 to 109.4] | 1.0 [0.8 to 1.1]

22. Secondary Outcome: Percentage of Participants Achieving Greater Than or Equal to 2-fold and 4-fold Increase From Before Vaccination (Baseline) in SARS-CoV-2 Anti-S1, Anti-RBD, and Anti-N Binding Antibody Levels
Time Frame: Day 56
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D
Number analyzed (Participants) | 114 | 115 | 117 | 116
percentage of participants
  Anti-N: >=2 Fold Increase From Baseline | 1.8 [0.2 to 6.2] | 2.6 [0.5 to 7.4] | 1.7 [0.2 to 6.0] | 2.6 [0.5 to 7.4]
  Anti-N: >=4 Fold Increase From Baseline | 0 [0.0 to 3.2] | 1.7 [0.2 to 6.1] | 0.9 [0.0 to 4.7] | 0 [0.0 to 3.1]
  Anti-RBD: >=2 Fold Increase From Baseline | 75.4 [66.5 to 83.0] | 96.5 [91.3 to 99.0] | 88.9 [81.7 to 93.9] | 3.4 [0.9 to 8.6]
  Anti-RBD: >=4 Fold Increase From Baseline | 64.0 [54.5 to 72.8] | 92.2 [85.7 to 96.4] | 84.6 [76.8 to 90.6] | 0.9 [0.0 to 4.7]
  Anti-S1: >=2 Fold Increase From Baseline | 90.4 [83.4 to 95.1] | 98.3 [93.9 to 99.8] | 95.7 [90.3 to 98.6] | 5.2 [1.9 to 10.9]
  Anti-S1: >=4 Fold Increase From Baseline | 85.1 [77.2 to 91.1] | 96.5 [91.3 to 99.0] | 92.3 [85.9 to 96.4] | 0.9 [0.0 to 4.7]

ADVERSE EVENTS:
Time Frame: Vaccination 1 and 2: Day 1 up to Day 207; Booster Vaccination: Day 208 to early termination (up to 396 days). Groups E-H1 also include participants who did not receive booster dose. As pre-specified, if a participant didn't receive booster dose but had safety data collected for the booster vaccination period, the participant was included in the placebo booster group for summarization (Group H1).
Description: Trt. A, B, C, D: Safety population. 1 participant in group A moved to group D in safety set due to not receiving correct dose. Trt. E1, F1, G1, H1: Booster Safety population. For Reactogenicity analysis, solicited AEs were documented by the participant in an eDiary, not assessed as serious or nonserious, and reported below in "Other" (Not Including Serious) Adverse Events.Unsolicited AEs are reported in Serious Adverse Events or "Other" (Not Including Serious) Adverse Events as assessed by PI.
Groups:
- Treatment A - Reactogenicity Analysis: Participants in this group received ARCT-021 7.5 mcg at Day 0 and placebo matched to ARCT-021 at Day 28. Participants who did not otherwise have any contraindications to additional study vaccinations were randomly assigned to ARCT-021, ARCT-154, ARCT-165, or placebo for a third (booster) dose of study vaccine given at Day 208.
- Treatment B - Reactogenicity Analysis: Participants in this group received ARCT-021 5 mcg at Day 0 and ARCT-021 5 mcg at Day 28. Participants who did not otherwise have any contraindications to additional study vaccinations were randomly assigned to ARCT-021, ARCT-154, ARCT-165, or placebo for a third (booster) dose of study vaccine given at Day 208.
- Treatment C - Reactogenicity Analysis: Participants in this group received ARCT-021 7.5 mcg at Day 0 and ARCT-021 7.5 mcg at Day 28. Participants who did not otherwise have any contraindications to additional study vaccinations were randomly assigned to ARCT-021, ARCT-154, ARCT-165, or placebo for a third (booster) dose of study vaccine given at Day 208.
- Treatment D - Reactogenicity Analysis: Participants in this group received placebo matched to ARCT-021 at Day 0 and placebo matched to ARCT-021 at Day 28. Participants who did not otherwise have any contraindications to additional study vaccinations were randomly assigned to ARCT-021, ARCT-154, ARCT-165, or placebo for a third (booster) dose of study vaccine given at Day 208.
- Treatment E1 - Reactogenicity Analysis: Participants in this group received booster dose of ARCT-021 5 mcg at Day 208.
- Treatment F1- Reactogenicity Analysis: Participants in this group received booster dose of ARCT-154 5 mcg at Day 208.
- Treatment G1 - Reactogenicity Analysis: Participants in this group received booster dose of ARCT-165 5 mcg at Day 208.
- Treatment H1 - Reactogenicity Analysis: Participants in this group received placebo at Day 208.
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E1 | Treatment F1 | Treatment G1 | Treatment H1 | Treatment A - Reactogenicity Analysis | Treatment B - Reactogenicity Analysis | Treatment C - Reactogenicity Analysis | Treatment D - Reactogenicity Analysis | Treatment E1 - Reactogenicity Analysis | Treatment F1- Reactogenicity Analysis | Treatment G1 - Reactogenicity Analysis | Treatment H1 - Reactogenicity Analysis
All-Cause Mortality (participants affected / at risk) | 0/145 | 0/144 | 0/145 | 0/146 | 0/44 | 0/41 | 0/42 | 0/99 | 0/142 | 0/142 | 0/144 | 0/146 | 0/43 | 0/38 | 0/38 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/145 | 3/144 | 1/145 | 3/146 | 0/44 | 0/41 | 1/42 | 0/99 | 0/142 | 0/142 | 0/144 | 0/146 | 0/43 | 0/38 | 0/38 | 0/39
Other Adverse Events (participants affected / at risk) | 49/145 | 15/144 | 27/145 | 11/146 | 10/44 | 9/41 | 11/42 | 19/99 | 113/142 | 107/142 | 120/144 | 30/146 | 35/43 | 25/38 | 28/38 | 10/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=145) | Treatment B (N=144) | Treatment C (N=145) | Treatment D (N=146) | Treatment E1 (N=44) | Treatment F1 (N=41) | Treatment G1 (N=42) | Treatment H1 (N=99) | Treatment A - Reactogenicity Analysis (N=142) | Treatment B - Reactogenicity Analysis (N=142) | Treatment C - Reactogenicity Analysis (N=144) | Treatment D - Reactogenicity Analysis (N=146) | Treatment E1 - Reactogenicity Analysis (N=43) | Treatment F1- Reactogenicity Analysis (N=38) | Treatment G1 - Reactogenicity Analysis (N=38) | Treatment H1 - Reactogenicity Analysis (N=39)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug abuse (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary venous thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=145) | Treatment B (N=144) | Treatment C (N=145) | Treatment D (N=146) | Treatment E1 (N=44) | Treatment F1 (N=41) | Treatment G1 (N=42) | Treatment H1 (N=99) | Treatment A - Reactogenicity Analysis (N=142) | Treatment B - Reactogenicity Analysis (N=142) | Treatment C - Reactogenicity Analysis (N=144) | Treatment D - Reactogenicity Analysis (N=146) | Treatment E1 - Reactogenicity Analysis (N=43) | Treatment F1- Reactogenicity Analysis (N=38) | Treatment G1 - Reactogenicity Analysis (N=38) | Treatment H1 - Reactogenicity Analysis (N=39)
COVID-19 (Infections and infestations) | 7 | 4 | 11 | 3 | 6 | 5 | 5 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 7 | 1 | 2 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 5 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asymptomatic COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 2 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 6 | 2 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 4 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immunisation reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 75 | 69 | 83 | 12 | 0 | 0 | 0 | 0 — Data reported for Vaccination 1.
Injection site Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 43 | 61 | 8 | 0 | 0 | 0 | 0 — Data reported for Vaccination 2.
Injection site Erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 28 | 16 | 11 | 0 | 0 | 0 | 0 — Data reported for Vaccination 1.
Injection site Erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 19 | 11 | 12 | 0 | 0 | 0 | 0 — Data reported for Vaccination 2.
Injection site Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 22 | 13 | 8 | 0 | 0 | 0 | 0 — Data Reported for Vaccination 1.
Injection site Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 15 | 6 | 4 | 0 | 0 | 0 | 0 — Data reported for Vaccination 2.
Injection site tenderness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 113 | 107 | 120 | 29 | 0 | 0 | 0 | 0 — Data reported for Vaccination 1.
Injection site tenderness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 88 | 103 | 21 | 0 | 0 | 0 | 0 — Data reported for Vaccination 2.
Injection site Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 22 | 14 | 15 | 2 — Data reported for Booster vaccination.
Injection site Erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 3 | 1 — Data reported for Booster Vaccination.
Injection site Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 3 | 0 — Data reported for Booster Vaccination.
Injection site tenderness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 25 | 28 | 5 — Data reported for Booster vaccination.
Fever (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 4 | 0 | 0 | 0 | 0 | 0 — Data Reported for Vaccination 1.
Fever (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 9 | 0 | 0 | 0 | 0 | 0 — Data reported for Vaccination 2.
Fever (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 2 | 1 — Data reported for Booster vaccination.
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 61 | 49 | 57 | 28 | 0 | 0 | 0 | 0 — Data reported for Vaccination 1.
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 39 | 56 | 22 | 0 | 0 | 0 | 0 — Data reported for Vaccination 2.
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 13 | 12 | 10 — Data reported for Booster vaccination.
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 67 | 52 | 58 | 30 | 0 | 0 | 0 | 0 — Data reported for Vaccination 1.
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 43 | 61 | 29 | 0 | 0 | 0 | 0 — Data reported for Vaccination 2.
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 30 | 13 | 19 | 10 — Data reported for Booster vaccination.
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 63 | 41 | 57 | 12 | 0 | 0 | 0 | 0 — Data reported for Vaccination 1.
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 45 | 45 | 19 | 0 | 0 | 0 | 0 — Data reported for Vaccination 2.
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 27 | 12 | 16 | 5 — Data reported for Booster vaccination.
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 30 | 22 | 25 | 12 | 0 | 0 | 0 | 0 — Data reported for Vaccination 1.
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 22 | 33 | 13 | 0 | 0 | 0 | 0 — Data reported for Vaccination 2.
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 8 | 12 | 5 — Data reported for Booster vaccination.
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 12 | 9 | 11 | 0 | 0 | 0 | 0 — Data reported for Vaccination 1.
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 9 | 12 | 7 | 0 | 0 | 0 | 0 — Data reported for Vaccination 2.
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 3 | 4 | 1 — Data reported for Booster vaccination.
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41 | 24 | 33 | 3 | 0 | 0 | 0 | 0 — Data reported for Vaccination 1.
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 17 | 31 | 7 | 0 | 0 | 0 | 0 — Data reported for Vaccination 2.
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 7 | 8 | 3 — Data reported for Booster vaccination.
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 18 | 23 | 14 | 0 | 0 | 0 | 0 — Data reported for Vaccination 1.
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 13 | 15 | 17 | 0 | 0 | 0 | 0 — Data reported for Vaccination 2.
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 7 | 4 | 4 — Data reported for Booster vaccination.
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 14 | 13 | 13 | 0 | 0 | 0 | 0 — Data reported for Vaccination 1.
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 6 | 24 | 9 | 0 | 0 | 0 | 0 — Data reported for Vaccination 2.
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 4 | 4 | 1 — Data reported for Booster vaccination.
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 — Data reported for Booster vaccination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT04668339/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT04668339/SAP_001.pdf